CLINICAL TRIAL: NCT01151631
Title: Occipital Nerve Stimulation in Medically Intractable Chronic Cluster Headache
Acronym: ICON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); Erasmus Medical Center (Other); Technical University of Twente (Other); Canisius-Wilhelmina Hospital (Other); University of Copenhagen (Other); University Hospital, Ghent (Other); Royal Free Hospital NHS Foundation Trust (Other); Medtronic (Industry); Centre Hospitalier Régional de la Citadelle (Other); Schmerzklinik Kiel (Unknown); University Hospital Schleswig-Holstein (Other); National Institute of Neuroscience, Budapest (Unknown)
Responsible Party: Principal Investigator, MDFerrari, Prof. M.D. Ferrari, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICON-01
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100% occipital nerve stimulation (Active Comparator): Stimulation frequency and pulse width will be uniformly held constant at 60 Hz and pulse width at 450 ms. The perception and discomfort amplitude will be defined by increasing the stimulation amplitude in steps of 0.1 V. The amplitude at which the patient starts feeling paraesthesis is called the perception threshold. The threshold at which the patient does not want the voltage to be increased any further because of painful sensations is designated the discomfort threshold. 100% stimulation is defined as stimulation at 90% of the range between perception and discomfort thresholds.
  Interventions: Device: occipital nerve stimulation
- 30% occipital nerve stimulation (Sham Comparator): 30% stimulation means a stimulation level at 30% of the range between perception threshold and 100% stimulation level
  Interventions: Device: occipital nerve stimulation

INTERVENTIONS:
Device: occipital nerve stimulation — Low occipital bilateral Quad Plus, midline to laterally directed, secured by titan anchors, connected to Versitrel. No trial stimulation. Suggested stimulation parameters: Pulse width: 450, Amplitude: protocol, Rate: 60
  Other Names: Versitrel™, Pisces Quad® Plus, Versitrel™ Patient Programmer

SUMMARY:
Cluster headache (CH) is a primary headache disorder characterized by recurrent short-lasting attacks (15 to 180 minutes) of excruciating unilateral periorbital pain accompanied by ipsilateral cranial autonomic signs. The 1-year prevalence of CH is about 0.1 %, the male: female ratio is 3:1. The majority of patients have cluster periods of weeks to months with frequent attacks which are alternated with symptom-free periods of months to several years; the episodic from of CH. In about 10% of patients the CH is chronic (CCH) in which either no remission occurs within 1 year or the remissions last less than 1 month. At least 10 % of CCH patients are refractory to medical treatment or cannot tolerate the treatments.

Recent pilot studies suggest that occipital nerve stimulation (ONS) in medically intractable CCH (MICCH) might offer an effective alternative to medical treatment. There are no randomised clinical trials and a placebo effect cannot be excluded. Long term tolerability is known from other indications.

Here the investigators propose a prospective, randomised, double blind, parallel group multi-centre international clinical study to compare the reduction in attack frequency from baseline of occipital nerve stimulation (ONS) in patients with MICCH between two different stimulation conditions: high (100%) and low (30%) stimulation.

Following implantation there will first be a run-in phase of 10 days of 10% stimulation intensity, followed by a stepwise monthly increase up to either 30% or 100%. Patients will be assessed monthly by a blinded assessor. The primary outcome measure is the mean number of attacks over the last 4 weeks of the double blind 6 month treatment period in the 100% versus the 30% treatment group. Hereafter, in an open extension phase of 6 months, all patients will receive 100% stimulation or the stimulation considered optimal by the patient.

Secondary outcome measures include the rate of responders (≥ 50% reduction in attack frequency during the last 4 weeks of each treatment period), patient's satisfaction, medication use, quality of life, mean pain intensity, economic evaluation and whether patients would recommend the treatment to another patient. The investigators will also investigate whether predictive factors can be identified for efficacy.

DETAILED DESCRIPTION:
Trigeminal autonomic cephalalgias (TACs) are characterized by frequent, short-lasting attacks of unilateral extremely severe headaches accompanied by ipsilateral facial autonomic features and are the most severe of the primary headache disorders. TACs include cluster headache (CH), paroxysmal hemicrania (PH) and short-lasting unilateral neuralgiform headache with conjunctival injection and tearing (SUNCT). CH is the most common form of TAC. The 1-year prevalence is about 1 in 1000, with the vast majority of patients having episodic CH (ECH): periods of weeks to months with frequent attacks which are alternated with symptom-free periods of several months to years. About 10% have chronic CH (CCH): attack free periods of less than one month in every 12 months, unless treatment is given. The chronic form can be primary unremitting from onset, or can be secondary, transform from the episodic form. CCH may spontaneously become episodic.

Effective acute treatments for CH attacks are injectable or intranasal triptans and oxygen inhalation. Steroids (only for a short period), verapamil, lithium carbonate and methysergide are the most effective preventive therapies. At least 10% of patients with CCH is or may become refractory to or cannot tolerate medical therapy. For patients with medically intractable CCH (MICCH) there is no common treatment. Different experimental treatments, such as deep brain stimulation (DBS), radiofrequency lesions, glycerol injections, gamma knife, and surgery or root section of the trigeminal nerve are either substantially ineffective, or have significant short-comings with serious complications such as death or neurological deficits such as anaesthesia dolorosa or lack of efficacy.

CH has considerable impact on socio-economic and personal functions due to direct costs of healthcare services and indirect costs of lost work days and decreased work efficacy. Higher pain scores and a higher percentage of patients with poor health due to pain and social functioning are found among CH patients compared with patients suffering from migraine. The impact on social functions, quality of life and use of healthcare of patients with MICCH is most likely even larger, although precise figures are not available. In the study of Burns et al. patients, suffering from MICCH, had on average over four attacks per day. Attacks of CH have been described by patients as being worse than child birth. Recently treatment of headache was listed as one of the top priorities of US National the Institute of Medicine's agenda for comparative-effectiveness research.

Functional imaging studies in CH identified activations in the region of the posterior hypothalamus, which led to the use of neurostimulation therapy in MICCH. Hypothalamic DBS was shown to be effective in some patients with MICCH but unfortunately this treatment is associated with a high risk of (even lethal) consequences.

Structures in the occipital region of the head are mainly innervated by the greater occipital nerve that is a branch of the C2 spinal root. Convergence of cervical, somatic trigeminal and dural trigeminovascular afferents on second order nociceptors in the brain stem is well documented. Stimulation of the greater occipital nerve increased metabolic activity in cervical regions of the spinal cord and in the trigeminal nucleus caudalis in the cat. In humans an occipital nerve blockade decreased the ipsi- and contralateral R2 response, confirming the anatomic and functional convergence of afferent cervical and trigeminal pathways. These studies suggest that modulation of these pathways may influence headache.

Suboccipital injection of corticosteroid with local anaesthetics was shown to be effective in a placebo-controlled trial. In this study 4 patients suffering from CCH were included. In all patients the attacks recurred eventually. The authors suggest that suboccipital steroid injections ought to be tried as a single shot treatment before invasive treatments are considered such as DBS, but in later studies this turned out to be of no predictive value of the response to neuromodulation therapies.

Along the same line, stimulation of the greater occipital nerve (ONS) has been tried with some success in intractable headaches including CCH. Burns et al. described 14 patients suffering from MICCH and were treated with ONS in an open retrospective study. Ten patients improved; three improved by 90% or more, 3 by 40%-90% and 4 by 20-30%. In a prospective open ONS study on MICCH patients Magis et al. showed a reduction in attack frequency of 79.9%. No serious complications were described in both studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of patients with CH shall be in accordance with The International Classification of Headache Disorders, 2nd Edition:

A. At least 5 attacks fulfilling criteria B-D B. Severe or very severe unilateral orbital, supraorbital and/or temporal pain lasting 15-180 minutes if untreated

C. Headache is accompanied by at least 1 of the following:

1. ipsilateral conjunctival injection and/or lacrimation
2. ipsilateral nasal congestion and/or rhinorrhoea
3. ipsilateral eyelid oedema
4. ipsilateral forehead and facial sweating
5. ipsilateral miosis and/or ptosis
6. a sense of restlessness or agitation D. Attacks have a frequency from 1 every other day to 8 per day E. Not attributed to another disorder

   * Chronic cluster headache A. Attacks fulfilling criteria A-E for Cluster headache B. Attacks recur over >1 year without remission periods or with remission periods lasting <1 month
   * ICHD-II criteria for CCH (see above)
   * Minimum mean attack frequency of 4 attacks per week
   * Minimum age of 18 years old
   * Signed study specific informed consent form
   * Agreeing to refrain from starting new prophylactic CH medication, including steroids, or any other therapy aimed at CH and agrees to maintain existing prophylactic CH medication from 4 weeks before entering the baseline period throughout the duration of the double blind phase of the study. It is allowed to change the dose of prophylactic medication during the study based on the opinion of the treating medical specialist.
   * Availability during follow-up period
   * An MRI to exclude structural lesions potentially causing CCH.
   * Medically intractable (see below)

Definition medically intractable :

Failed adequate trials of regulatory approved and conventional treatments according to local national guidelines

Adequate trial:

Appropriate dose and duration of treatment according to local guidelines Appropriate length of time Consideration of medication overuse

Failed:

No therapeutic or unsatisfactory effect, intolerable side effects, contraindications to use

Must have tried agents of at least three classes of the following, of which 1 and 2 are obligatory, and 1 should come from 3-5: (recommendation of Goadsby et al. applied to Dutch national guidelines)

1. Verapamil
2. Lithium
3. Methysergide
4. Topiramate
5. Gabapentin

Exclusion Criteria:

* Other significant neurological or disabling diseases which in the opinion of the clinician may interfere with the study
* Pregnancy or the wish to become pregnant during the study period
* Cardiac pacemaker and other neuromodulatory devices
* Psychiatric or cognitive disorders and/or behavioural problems which in the opinion of the clinician may interfere with the study
* Taking CH prophylactic medication for conditions other than CH which in the opinion of the clinician may interfere with the study
* Serious drug habituation and/or overuse of acute headache medication for other headaches than CH
* Inability to complete the (electronic) diary in a sensible and accurate manner
* Structural intracranial or cervical vascular lesions that may potentially cause CH
* Previous destructive surgery involving the C2 or C3 roots (vertebrae) or deep brain stimulation
* Enrollment in other clinical studies that may confound the results of this study
* Requiring anticoagulation therapy or antithrombotic or thrombocyte aggregation-inhibitor for a concomitant condition that cannot be stopped peri-operatively. The local peri-operative protocol of each individual participating centre will be followed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-10; Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The mean attack frequency (MAF) over the last 4 weeks in the 100% and the 30% treatment groups | 6 months
  An attack is defined as any attack recognised by the patient as being a CH attack. So also the attacks treated with oxygen or triptans.

SECONDARY OUTCOMES:
The MAF during follow up | for each 4 week period of the whole follow-up period
The mean attack intensity (on a scale from 0-10) will be calculated and will be compared between and within the 2 groups. | over the last 4 weeks for each group at baseline, 6 and 12 months follow up
Rate of responders (>50% reduction in attack frequency in the last 4 weeks compared to baseline) will be calculated and compared between groups | 6 and 12 months follow up
Economic evaluation | baseline and 6 months follow-up
Anticipated group randomisation | at 12 months follow-up
Awareness of paraesthesias | weekly during 6 months follow up
The use of acute attack medication | during the last 4 weeks at baseline periode and 6 months follow up
Patient satisfaction | 6 and 12 months follow up
  The investigators will ask the patient whether he/she would recommend the treatment to another patient using a 5 point (Likert) scale: Strongly disagree, disagree, neither agree nor disagree, agree, strongly agree.
Responder identification | 12 months follow up
  It is also investigated whether predictive factors can be identified with respect to the outcome in a hypothesis generating manner. We will look at the body mass index (BMI) and assess the predictive value of response after 5-7 days.
Adverse events | 1 year
  All and treatment-related adverse events will be documented by the investigators.
MAF | 6 months
  MAF: We will repeat the primary analysis, with the MAF as outcome instead of the logarithm of the MAF.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ferrari, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (7):
- CHR La Citadelle hospital, Liège, Belgium
- Schmerzklinik Kiel, Kiel, Germany
- National Institute of Neuroscience, Budapest, Hungary
- Netherlands (4):
  - Boerhaave MC, Amsterdam
  - Atrium medical centre, Heerlen
  - Leiden University Medical Center, Leiden
  - Canisius Wilhelmina Hospital, Nijmegen

REFERENCES:
- [Background] Burns B, Watkins L, Goadsby PJ. Treatment of intractable chronic cluster headache by occipital nerve stimulation in 14 patients. Neurology. 2009 Jan 27;72(4):341-5. doi: 10.1212/01.wnl.0000341279.17344.c9. PMID 19171831
- [Background] Burns B, Watkins L, Goadsby PJ. Treatment of medically intractable cluster headache by occipital nerve stimulation: long-term follow-up of eight patients. Lancet. 2007 Mar 31;369(9567):1099-106. doi: 10.1016/S0140-6736(07)60328-6. PMID 17398309
- [Background] Magis D, Allena M, Bolla M, De Pasqua V, Remacle JM, Schoenen J. Occipital nerve stimulation for drug-resistant chronic cluster headache: a prospective pilot study. Lancet Neurol. 2007 Apr;6(4):314-21. doi: 10.1016/S1474-4422(07)70058-3. PMID 17362835
- [Derived] Brandt RB, Mulleners W, Wilbrink LA, Brandt P, van Zwet EW, Huygen FJ, Ferrari MD, Fronczek R; ICON study group. Intra- and interindividual attack frequency variability of chronic cluster headache. Cephalalgia. 2023 Feb;43(2):3331024221139239. doi: 10.1177/03331024221139239. PMID 36739508
- [Derived] Wilbrink LA, de Coo IF, Doesborg PGG, Mulleners WM, Teernstra OPM, Bartels EC, Burger K, Wille F, van Dongen RTM, Kurt E, Spincemaille GH, Haan J, van Zwet EW, Huygen FJPM, Ferrari MD; ICON study group. Safety and efficacy of occipital nerve stimulation for attack prevention in medically intractable chronic cluster headache (ICON): a randomised, double-blind, multicentre, phase 3, electrical dose-controlled trial. Lancet Neurol. 2021 Jul;20(7):515-525. doi: 10.1016/S1474-4422(21)00101-0. PMID 34146510

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT01151631/Prot_SAP_000.pdf